CLINICAL TRIAL: NCT03673254
Title: A Prospective Multinational European Study on Evaluation of Practices and Prognostic Factors of Percutaneous Coronary Interventions (PCI) of Calcified Complex Lesions Using Rotational Atherectomy Device.
Brief Title: Evaluation of Practices and Prognostic Factors of Percutaneous Coronary Interventions (PCI) of Calcified Complex Lesions Using Rotational Atherectomy Device.
Acronym: Eurotaclub
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8373
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Angioplasty
Keywords: rotational atherectomy device,

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: rotational atherectomy device — angioplasty with rotational atherectomy device on a nonselected population

SUMMARY:
In spite of technological advances, PCI of complex calcified coronary lesions remain a challenge.

Observational studies demonstrate that moderate or severe calcifications in lesions to treat are associated with an increase in mortality, in myocardial infarctions, in stent thrombosis, and in complementary revascularizations. Rotational atherectomy is now part of therapeutic armamentarium of interventional cardiologists for the treatment of some complex calcified coronary lesions. Last recommendations of the European Society of Cardiology about revascularizations indicate that rotational atherectomy should be used for "the preparation of calcified or massive fibrotic lesions that cannot be crossed by a balloon or for an optimal dilatation before stenting". However, this technique is not frequently used and limited to high-volume PCI centers. Even though rotational atherectomy demonstrated an improvement in immediate success of complex lesions, the longterm reduction of cardiovascular events after active stenting has not been proved. In observational studies, the results are not consistent because of many selection biases that influence the choice of an angioplasty with rotational atherectomy device (calcifications, severity of the disease). Furthermore, this technique needs operators with a certain amount of experience. The fundamentals of an optimal use of rotational atherectomy remain to be defined (duration and speed of burr, anti-platelet treatments...).

ELIGIBILITY:
Inclusion Criteria:

* patients with angioplasty that requires the rotational atherectomy device
* agree to participate in this study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be included all patients who undergo an angioplasty that requires the rotational atherectomy device and who agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Determination of the prognostic impact of a myocardial | One year
  Composite safety endpoint collecting cardiovascular events (cardiovascular death, myocardial infarction, target lesion revascularization, stroke, stent thrombosis, coronary bypass)

SECONDARY OUTCOMES:
Frequency of angiographic complications for an optimization of PCI by rotational atherectomy | one year
  Number of angiographic complications
Frequency of in-hospital events | One year
  Number of in-hospital events

CONTACTS AND LOCATIONS:
Overall Officials: Didier CARRIE, MD, Principal Investigator — Univesity Hospital Toulouse
Locations (16):
- Hanush Krankenhaus, Vienna, Austria
- France (4):
  - La clinique des eaux claires, Grenoble
  - Les Nouvelles Cliniques Nantaises, Nantes
  - University Hospital Nimes, Nîmes
  - University Hospital Toulouse, Toulouse
- Augusta Krankenhaus, Düsseldorf, Germany
- St Luke's Hospital, Thessaloniki, Greece
- Italy (2):
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - University of Verona, Verona
- Poland (4):
  - University Hospital of Bialystok, Bialystok
  - Interventional Cardiology Clinic, Jagiellonina University, Krakow
  - University Hospital in Poznan, Poznan
  - Wojskowy Szpital Kliniczny Wroclaw, Wroclaw
- Moscow, Russia
- Spain (2):
  - Hospital Del mar, Barcelona
  - Hospital Universitario Central de la Defensa "Gomez Ulla", Madrid

IPD SHARING:
Plan to Share IPD: Undecided